CLINICAL TRIAL: NCT04804267
Title: A Randomized, Double-blinded, Placebo-controlled, Multicenter Study to Evaluate the Clinical Equivalence of Two Linaclotide Products and the Efficacy and Safety of the Test Formulation of Linaclotide in the Treatment of Chronic Idiopathic Constipation
Brief Title: Evaluation of Clinical Equivalence Between Two Linaclotide Products in the Treatment of Chronic Idiopathic Constipation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-20078-501
Record Dates: First submitted 2021-03-10; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-01

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Linaclotide Manufactured by Jiangsu Hansoh Pharmaceutical Co., Ltd. Drug: Linaclotide 145μg orally once daily
  Interventions: Drug: Linaclotide
- Active Comparator (Active Comparator): LINZESS® Manufactured by Almac Pharma Services Limited Drug: Linaclotide 145μg orally once daily
  Interventions: Drug: LINZESS®
- Placebo Comparator (Placebo Comparator): Placebo Drug: Placebo orally once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linaclotide — Manufactured by Jiangsu Hansoh Pharmaceutical Co., Ltd. Drug: Linaclotide 145μg orally once daily
  Arms: Experimental
Drug: LINZESS® — Manufactured by Almac Pharma Services Limited Drug: Linaclotide 145μg orally once daily
  Arms: Active Comparator
Drug: Placebo — Drug: Placebo orally once daily
  Arms: Placebo Comparator

SUMMARY:
The objective of this study is to evaluate the clinical equivalence of the test formulation of Linaclotide compared to the marketed formulation LINZESS® in patients with Chronic Idiopathic Constipation, and to evaluate the efficacy and safety of the test formulation of Linaclotide in the treatment of Chronic Idiopathic Constipation.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled, multicenter study to evaluate the clinical equivalence of the test formulation of Linaclotide (manufactured by Jiangsu Hansoh Pharmaceutical Co., Ltd.) compared to the marketed formulation LINZESS® in patients with Chronic Idiopathic Constipation.

ELIGIBILITY:
Inclusion Criteria:

* Males or nonpregnant females aged ≥ 18 years with a clinical diagnosis of chronic idiopathic constipation defined as < 3 spontaneous bowel movements (SBMs) per week and confirmed by daily diary during baseline period;

Have 1 or more of the following symptoms related to bowel movements for the past 3 months with symptom onset at least 6 months before screening and confirmed by daily diary during the 2-week baseline period:

* lumpy or hard stools for more than 25% of the bowel movements (Bristol Stool Form Scale 1 to 2)
* sensation of incomplete evacuation following more than 25% of the bowel movements
* straining at defecation more than 25% of the time Willing to discontinue any laxatives used before the Pretreatment Visit in favor of the protocol-defined Rescue Medicine; Agree to refrain from making any new major life-style changes that may have affected CIC symptoms; Females of child-bearing potential have a negative pregnancy test prior to beginning therapy and agree to use effective contraceptive methods during the study and until 30 days after the last dose; Males who have partners of childbearing potential agree to use effective contraceptive methods during the study and until 30 days after the last dose.

Exclusion Criteria:

* Meet the Rome IV criteria for Irritable Bowel Syndrome or the Rome IV criteria for Opioid-Induced Constipation; Have a potential central nervous system cause of constipation (e.g., Parkinson's disease, spinal cord injury, and multiple sclerosis, etc.); Have a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility; Subjects with documented mechanical bowel obstruction (e.g., bowel obstruction due to tumor, hernia), megacolon/megarectum, or diagnosis of pseudo-obstruction; Have ever had a fecal impaction that required hospitalization or emergency room treatment, or has a history of cathartic colon, laxative or enema abuse, ischemic colitis, or pelvic floor dysfunction (unless successful treatment has been documented by a normal balloon expulsion test); Subjects with known or suspected organic disorders of the large or small bowel (e.g., inflammatory bowel disease, ulcerative colitis, Crohn's Disease); Subjects with constipation secondary to a documented cause (e.g., surgery, bowel resection); Diagnosis or family history of familial adenomatous polyposis, hereditary nonpolyposis colorectal cancer, or any other form of familial colorectal cancer; Have a history of cancer other than treated basal cell or squamous cell carcinoma of the skin in the past 5 years; Have currently unexplained and clinically significant alarm symptoms (lower GI bleeding [rectal bleeding or heme-positive stool], anemia, weight loss) or systemic signs of infection or colitis; Have currently active peptic ulcer disease; Have a history of diabetic neuropathy; Have untreated hypothyroidism or treated hypothyroidism for which the dose of thyroid hormone has not been stable for at least 6 weeks at the time of the Screening Visit; Have a history of diverticulitis or any chronic condition (e.g., chronic pancreatitis, polycystic kidney disease, ovarian cysts, endometriosis) that can be associated with abdominal pain or discomfort and could confound the assessments in this trial; Have clinically significant cardiovascular, liver, lung, neurologic, renal or psychiatric disorder, or clinically significant laboratory abnormalities, ineligible to participate in the study as determined by the investigator; Have a history of drug or alcohol abuse in the past 12 months before screening; Bariatric surgery for treatment of obesity or surgery to remove a segment of the GI tract at any time before screening; any gastrointestinal or abdominal surgical procedure during the 3 months before screening; any other major surgery during the 30 days before screening; Use of systemic antibiotics within 4 weeks prior to enrolment; Unwilling or unable to abide by the restrictions regarding use of prohibited medicines; Have received any investigational drug during the 3 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
The number of spontaneous bowel movements (SBM) during Week 1 | 1 week

SECONDARY OUTCOMES:
Percentage of 12-Week complete spontaneous bowel movements (CSBMs) overall responders | 12 week
The number of CSBM during Week 1 compared to baseline | 1 week
The proportion of patients with a SBM within 24 hours of receiving the first dose | 24 hours after the first dose
Time to first SBM after the first dose | up to 1 week
The proportion of patients with 12-Week CSBM frequency rate (CSBMs/week) ≥3 | 12 week
Change from baseline in 12-Week CSBM frequency rate (CSBMs/week) | 12 week
Change from baseline in 12-Week SBM frequency rate (SBMs/week) | 12 week
Change From Baseline in 12-Week Stool Consistency Assessment (seven-point ordinal Bristol Stool Form Scale) | 12 week
Change From Baseline in 12-Week Severity of Straining Assessment (five-point ordinal scale) | 12 week
Change From Baseline in 12-Week Abdominal Discomfort Assessment (five-point ordinal scale) | 12 week
Change From Baseline in 12-Week Bloating Assessment (five-point ordinal scale) | 12 week
Change From Baseline in 12-Week Constipation Severity Assessment (five-point ordinal scale) | 12 week
Change From Baseline in PAC-QOL score (Patient Assessment of Constipation Quality of Life questionnaire) | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Medical Collge of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No